CLINICAL TRIAL: NCT04943432
Title: Open Trial of a Behavioral Activation Telepsychology Intervention for People Who Inject Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1458; 1F31DA049457 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-29 (Actual); Results first posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-08

CONDITIONS: Intravenous Drug Usage
Keywords: People who inject drugs; Behavioral Activation; Telepsychology; Psychosocial Treatment; Harm Reduction; Low-threshold
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People who inject drugs (Experimental): People who inject drugs recruited from a needle exchange program who will participate in a psychosocial intervention
  Interventions: Behavioral: Behavioral Activation

INTERVENTIONS:
Behavioral: Behavioral Activation — 8 sessions of harm reduction-focused Behavioral Activation for Substance Use

SUMMARY:
The study has two aims: 1) To examine the feasibility and acceptability of administering a telepsychology Behavioral Activation (BA) treatment for substance use among non-treatment-seeking people who inject drugs (PWID); 2) To test the initial efficacy of the treatment from pretreatment to a 1-month follow-up on substance-related problems, readiness to change drug use, and BA. The intervention is hypothesized to be feasible and well-accepted, and within-subject analyses are hypothesized to demonstrate decreases in substance-related problems and increases in readiness to change drug use and BA from pretreatment to a 1-month follow-up.

The study aims to recruit N=25 non-treatment-seeking PWID from a syringe exchange program (estimated treated sample n=15). Participants will receive 8 sessions of BA over 4 weeks, and assessment of study outcome measures will occur at pretreatment, post-treatment, and a one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Reports regular recent injection drug use (defined as injecting drugs on at least one day in the last week and injecting drugs for at least two months)
* Can identify at least one goal or area of change to address during treatment
* Has regular (at least twice weekly) access to an electronic device that can make phone or video calls and has access to the internet to complete online questionnaires

Exclusion Criteria:

* Attending or on a wait list to receive psychosocial substance use treatment
* <5th grade reading level
* Impairment due to active psychosis
* Unable to give informed, voluntary, written consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Paquette, MPS, MA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | People Who Inject Drugs
Started | 23
Received Intervention | 19
Completed | 17
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: Participants who completed the pretreatment assessment and enrolled in the study.
Groups:
- People Who Inject Drugs: People who inject drugs recruited from a needle exchange program who will participate in a psychosocial intervention. Behavioral Activation: 8 sessions of harm reduction-focused Behavioral Activation for Substance Use
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Behavioral Activation Assessed With Behavioral Activation for Depression Scale (BADS) Score
Description: Behavioral Activation for Depression Scale (BADS) total score; Scale range 0-150, higher scores indicate greater activation (positive outcome).
Time Frame: pretreatment (T1), immediately after (or up to 2 weeks after) treatment completion (T2), and 1 month (or up to 2 months) posttreatment (T3), where average treatment duration was 4 weeks
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 22
score on a scale
  T1 | 77.00 (28.93)
  T2: number analyzed (Participants) | 16
  T2 | 86.75 (36.12)
  T3: number analyzed (Participants) | 9
  T3 | 69.67 (17.99)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2 - T1; Test type: Superiority; p = 0.06, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3 - T1; Test type: Superiority; p = 0.68, t-test, 2 sided

2. Primary Outcome: Change in Substance Use Problem Recognition Score Assessed With Recognition Subscale of Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) Score (Readiness to Change Drug Use)
Description: Outcome is subscale score on Recognition subscale of Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES); Range of 7-35, higher scores indicate greater problem recognition.
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 22
score on a scale
  T1 | 28.82 (4.80)
  T2: number analyzed (Participants) | 16
  T2 | 30.25 (4.04)
  T3: number analyzed (Participants) | 10
  T3 | 29.17 (4.44)

3. Primary Outcome: Change in Taking Steps to Change Substance Use Assessed With Taking Steps Subscale of Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) Score (Readiness to Change Drug Use)
Description: Outcome is subscale score on Taking Steps subscale of Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES); Range of 8-40, higher scores indicate greater steps to change (positive outcome)
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 22
score on a scale
  T1 | 26.28 (6.77)
  T2: number analyzed (Participants) | 16
  T2 | 32.62 (6.39)
  T3: number analyzed (Participants) | 10
  T3 | 29.91 (6.60)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2-T1; Test type: Superiority; p = .01, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3-T1; Test type: Superiority; p = .32, t-test, 2 sided

4. Primary Outcome: Change in Substance-related Problems Assessed With Short Inventory of Problems - Alcohol and Drugs (SIP) Score
Description: Short Inventory of Problems - Alcohol and Drugs (SIP) total score; Scale range 0-45, higher scores indicate greater problems (negative outcome)
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 23
score on a scale
  T1 | 22.92 (11.90)
  T2: number analyzed (Participants) | 16
  T2 | 22.08 (12.55)
  T3: number analyzed (Participants) | 8
  T3 | 33.34 (11.22)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2-T1; Test type: Superiority; p = .44, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3-T1; Test type: Superiority; p = .007, t-test, 2 sided

5. Primary Outcome: Treatment Attendance (Feasibility)
Description: Number of treatment sessions attended; Range 0-8; Higher number indicates greater attendance (positive outcome)
Time Frame: During the intervention, or up to 6 weeks after the pretreatment assessment, where average treatment duration was 4 weeks
Population: All participants who enrolled in the study
Measure: Mean (Standard Deviation); unit: Treatment sessions attended
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 23
Treatment sessions attended
  All participants | 4.5 (3.4)
  Participants who attended at least one session: number analyzed (Participants) | 19
  Participants who attended at least one session | 5.5 (2.9)

6. Primary Outcome: Treatment Satisfaction Assessed With Client Satisfaction Questionnaire Score (Acceptability)
Description: Client Satisfaction Questionnaire; Scale range 8 to 32, higher scores indicate greater satisfaction (positive outcome)
Time Frame: At the Posttreatment assessment (T2), which occurs after treatment completion or a maximum of 8 weeks after the pretreatment assessment, where average treatment duration was 4 weeks
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 15
score on a scale | 28.9 (3.0)

7. Primary Outcome: Therapeutic Alliance Assessed With Working Alliance Inventory Score (Acceptability)
Description: Outcome is mean of all items on Working Alliance Inventory; Range 1-5, higher scores indicate greater therapeutic alliance (positive outcome)
Time Frame: as for outcome 6
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 15
score on a scale | 4.5 (0.5)

8. Secondary Outcome: Change in Depressive Symptoms Assessed With Patient Health Questionnaire 9 (PHQ-9 Depression) Score
Description: Patient Health Questionnaire 9 (PHQ-9 Depression); Scale range 0-27, higher scores indicate greater depressive symptoms (negative outcome)
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 23
score on a scale
  T1 | 14.17 (9.54)
  T2: number analyzed (Participants) | 16
  T2 | 11.73 (9.37)
  T3: number analyzed (Participants) | 9
  T3 | 15.14 (8.07)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2-T1; Test type: Superiority; p = .01, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3-T1; Test type: Superiority; p = .11, t-test, 2 sided

9. Secondary Outcome: Change in Anxiety Symptoms Assessed With General Anxiety Disorder-7 (GAD-7 Anxiety) Score
Description: General Anxiety Disorder-7 (GAD-7 Anxiety); Scale range 0-21, higher scores indicate greater anxiety symptoms (negative outcome)
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 22
score on a scale
  T1 | 10.14 (7.46)
  T2: number analyzed (Participants) | 16
  T2 | 11.31 (6.86)
  T3: number analyzed (Participants) | 9
  T3 | 11.22 (7.56)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2-T1; Test type: Superiority; p = .82, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3-T1; Test type: Superiority; p = .36, t-test, 2 sided

10. Secondary Outcome: Change in HIV Risk Behaviors Assessed With HIV Risk Behavior Scale (HRBS) Score
Description: HIV Risk Behavior Scale (HRBS); Scale range 0-55, higher scores indicate greater HIV risk behavior (negative outcome)
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 23
score on a scale
  T1 | 16.61 (6.20)
  T2: number analyzed (Participants) | 16
  T2 | 13.25 (7.78)
  T3: number analyzed (Participants) | 9
  T3 | 8.00 (5.52)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2-T1; Test type: Superiority; p = .34, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3-T1; Test type: Superiority; p = .02, t-test, 2 sided

11. Secondary Outcome: Change in Substance Use Risk Assessed With Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) Score
Description: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST); Scale range 0-44, higher scores indicate greater substance use risk (negative outcome)
Time Frame: from Pretreatment up to 2 months posttreatment
Population: Results are not available for this outcome due to a survey programming error resulting in invalid data for the ASSIST.
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Substance Use Frequency Assessed With Timeline Followback (TLFB) Interview
Description: Percent days with any substance use, assessed via Timeline followback (TLFB) Interview; Range 0-100%, higher scores indicate greater substance use frequency (negative outcome)
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 22
percentage of days
  T1 | 95.46 (8.27)
  T2: number analyzed (Participants) | 16
  T2 | 85.28 (27.47)
  T3: number analyzed (Participants) | 10
  T3 | 85.13 (31.59)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2-T1; Test type: Superiority; p = .14, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3-T1; Test type: Superiority; p = .29, t-test, 2 sided

13. Secondary Outcome: Goal Attainment Assessed With Modified Goal Attainment Scale Score
Description: Modified Goal Attainment Scale; Range 0-5, higher scores indicate greater goal attainment (positive outcome)
Time Frame: During the intervention, or up to 6 weeks after the baseline assessment, where average treatment duration was 4 weeks
Population: This outcome measure was dropped (never added to the survey) as it was not one of the primary or secondary outcomes delineated in the study protocol. Data for this measure were not collected.
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 0

14. Secondary Outcome: Environmental Reward Assessed With Environmental Reward Observation Scale (EROS) Score
Description: Environmental Reward Observation Scale (EROS); Scale range 10-40, higher scores indicate greater environmental reward (positive outcome)
Time Frame: as for outcome 1
Population: Data are included for all participants who provided valid assessment data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | People Who Inject Drugs
Number analyzed (Participants) | 16
score on a scale
  T1 | 22.50 (6.52)
  T2: number analyzed (Participants) | 10
  T2 | 28.0 (5.79)
  T3: number analyzed (Participants) | 10
  T3 | 22.80 (6.53)
Statistical Analysis 1: Comparison: People Who Inject Drugs; T2-T1; Test type: Superiority; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: People Who Inject Drugs; T3-T1; Test type: Superiority; p = .23, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From the time of informed consent through the 1-month follow-up assessment, a period of up to 3 months (where average duration was approximately 2 months).
Arm/Group | People Who Inject Drugs
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04943432/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04943432/ICF_000.pdf